CLINICAL TRIAL: NCT06873945
Title: A PHASE 3, EXTERNAL AND SYNTHETIC PLACEBO-CONTROLLED RANDOMIZED STUDY WITH DOSE-UP FOR NON-RESPONDERS TO INVESTIGATE SAFETY AND EFFICACY OF RITLECITINIB 50 MG AND 100 MG ONCE DAILY IN ADULT AND ADOLESCENT PARTICIPANTS 12 YEARS OF AGE AND OLDER WITH ALOPECIA AREATA
Brief Title: A Study of 2 Doses of Ritlecitinib in People 12 Years of Age and Older With Alopecia Areata
Acronym: ALLEGRO-100
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7981094; 2024-519370-40-00 (Registry Identifier: CTIS (EU))
Expanded Access: NCT05522556 (Available)
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Alopecia Areata
Keywords: alopecia universalis; alopecia totalis; alopecia; patchy hair loss; diffuse hair loss; ophiasis; hair disease; Ritlecitinib; Litfulo; hair loss; adolescents; adults
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis; Alopecia; Hair Diseases | interventions — PF-06651600

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ritlecitinib 100 mg (Experimental): Randomized to Ritlecitinib 100 mg QD for 48 weeks. In addition to the active Ritlecitinib 100 mg capsule, a placebo capsule matching the Ritlecitinib 50 mg capsule will be given in order to maintain the blind.
  Interventions: Drug: Ritlecitinib 100 mg; Drug: Placebo - 50 mg
- Ritlecitinib 50 mg (Experimental): Randomized to Ritlecitinib 50 mg QD for 24 weeks. Depending on response status at Week 24 (ie, whether the participant has a SALT score of less than or equal to 20), the participant may be re-randomized to Ritlecitinib 50 mg QD or Ritlecitinib 100 mg QD for another 24 weeks.
  In addition to the active Ritlecitinib 50 mg capsule, a placebo capsule matching the Ritlecitinib 100 mg capsule will be given in order to maintain the blind.
  Interventions: Drug: Ritlecitinib 50 mg; Drug: Placebo - 100 mg
- External Placebo (No Intervention): This group will be constructed using participant-level data at Week 24 from placebo groups of the appropriately chosen Pfizer clinical studies of Ritlecitinib in participants with alopecia areata. This data will be used for comparison between each Ritlecitinib dose and placebo at Week 24.
  As this arm will utilize data from other studies, no participants will be randomized to receive only placebo in this study.
- Synthetic Placebo (No Intervention): This group will be constructed using participant-level data up to Week 36 from the placebo groups of the appropriately chosen Pfizer clinical studies of Ritlecitinib in participants with alopecia areata and a longitudinal model and extrapolation. This data will be used for comparison between Ritlecitinib 100 mg and placebo at Week 36.
  As this arm will utilize data from other studies, no participants will be randomized to receive only placebo in this study.

INTERVENTIONS:
Drug: Ritlecitinib 100 mg — 100 mg Capsule
  Other Names: PF-06651600; Litfulo
  Arms: Ritlecitinib 100 mg
Drug: Ritlecitinib 50 mg — 50 mg Capsule
  Other Names: PF-06651600; Litfulo
  Arms: Ritlecitinib 50 mg
Drug: Placebo - 100 mg — Capsule (to match Ritlecitinib 100 mg)
  Arms: Ritlecitinib 50 mg
Drug: Placebo - 50 mg — Capsule (to match Ritlecitinib 50 mg)
  Arms: Ritlecitinib 100 mg

SUMMARY:
The purpose of the study is to learn about the safety and effects of the study medicine (called ritlecitinib) for the treatment of alopecia areata. Alopecia areata is a disease that causes hair loss on the scalp, face, and areas of the body.

Ritlecitinib is approved in many countries at a dose of 50 mg (milligram) taken by mouth once a day for the treatment of patients 12 years and older with severe alopecia areata. This study will look at both the 50 mg dose and a 100 mg dose.

This study is seeking participants who:

* Are 12 years of age or older
* Have a diagnosis of alopecia areata
* Have lost 50% or more of the hair on their scalp
* Do not have any other conditions that causes hair loss
* Are willing to stop all other treatments that they may be taking for alopecia areata

About 550 participants will take part in in this study.

Participants will be chosen by chance, like drawing names out of a hat, to receive 1 of 2 different amounts of ritlecitinib (50 mg and 100 mg) taken by mouth once daily.

The 2 doses of ritlecitinib in this study will be compared to each other and also to data from previous studies. This will help to see if the 100 mg dose of ritlecitinib is safe and effective.

People will be in this study for about 13 months. During the study, participants will need to visit the study site up to 9 times. Participants will undergo various tests and procedures such as:

* alopecia areata assessment,
* physical examinations,
* hearing tests,
* blood tests,
* x-ray,
* ECG (electrocardiogram),
* photographs of the scalp and eyes. Participants will also be asked to complete questionnaires about their alopecia areata.

ELIGIBILITY:
Inclusion Criteria:

Age:

1. 18 years of age or older at screening. Adolescents (12 to <18 years of age at screening) are also eligible for this study, but only if permitted by the local IRB/EC and local regulatory health authority (if applicable). Where these approvals have not been granted, only participants 18 years of age and older at screening will be enrolled.

   Disease Characteristics:
2. Must meet the following alopecia areata criteria at both Screening and Baseline:

   1. Have a clinical diagnosis of alopecia areata with no other etiology of hair loss.
   2. ≥50% hair loss of the scalp, as measured by SALT, without evidence of terminal hair regrowth within the previous 6 months.
   3. Current episode of hair loss ≤10 years.

Exclusion Criteria:

Medical Conditions:

1. Diseases or conditions other than alopecia areata which affect hair loss, including other types of alopecia, other scalp disease that may impact the alopecia areata assessment, or active systemic diseases that may cause hair loss.
2. History of severe allergic or anaphylactoid reaction to any kinase inhibitor or a known allergy/hypersensitivity to any component (including excipients) of the study intervention.
3. Any psychiatric condition including recent or active suicidal ideation or behavior that meets protocol-defined criteria.
4. General Infection History:

   * Have a history of systemic infection requiring hospitalization or parenteral therapy (antimicrobial, antiviral, antiparasitic, antiprotozoal, or antifungal), or as otherwise judged clinically significant by the investigator, within 3 months prior to Day 1.
   * Have active acute or chronic infection requiring treatment with oral antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks prior to Day 1. NOTE: participants may be rescreened after the infection resolves.
   * Evidence or history of untreated, currently treated or inadequately treated active or latent infection with Mycobacterium tuberculosis.
5. Specific Viral Infection History:

   * History (single episode) of disseminated herpes zoster or disseminated herpes simplex, or a recurrent (more than one episode of) localized, dermatomal herpes zoster.
   * Infected with hepatitis B or hepatitis C viruses: all participants will undergo screening for hepatitis B and C for eligibility.
6. Other Medical Conditions:

   * Have hearing loss with progression over the previous 5 years, sudden hearing loss, or middle or inner ear disease such as otitis media, cholesteatoma, Meniere's disease, labyrinthitis, or other auditory condition that is considered acute, fluctuating or progressive.
   * Abnormal findings on the screening chest imaging (eg, chest x-ray) including, but not limited to, presence of active TB or other infections, cardiomyopathy, or malignancy. Chest imaging may be performed up to 12 weeks prior to Screening.
   * Have any malignancies or have a history of malignancies with the exception of adequately treated or excised nonmetastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
   * Have a history of any lymphoproliferative disorder such as EBV-related lymphoproliferative disorder, history of lymphoma, history of leukemia, or signs and symptoms suggestive of current lymphatic or lymphoid disease.
   * Significant trauma or major surgery within 1 month of the first dose of study drug or considered in imminent need for surgery.
7. Adolescent participants 12 to <18 years of age without one of the following:

   * Documented evidence from a health professional of having received varicella vaccination (2 doses); or
   * Evidence of prior exposure to varicella zoster virus (VZV) based on serological testing (ie, a positive VZV IgG Ab result) at Screening.
8. Any medical or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

   Prior/Concomitant Therapy:
9. Current or prior use of any prohibited medication(s), vaccine(s), or treatment(s) within the protocol-defined timelines.

   Prior/Concurrent Clinical Study Experience:
10. Previous administration with an investigational drug or vaccine within 8 weeks (or longer as determined by the local requirement) or 5 half-lives (whichever is longer) before the first dose of study intervention in this study. Participation in studies of other investigational products (drug or vaccine) at any time during their participation in this study.

    Diagnostic Assessments:
11. Any exclusionary abnormalities in laboratory values at Screening, as assessed by the study-specific laboratory and, if deemed necessary, confirmed by a single repeat.
12. Screening standard 12-lead ECG that demonstrates clinically relevant abnormalities.

    Other Exclusion Criteria:
13. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-03-09 (Estimated); Study Completion 2027-03-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with absolute Severity of Alopecia Tool (SALT) score less than or equal to 20 | Week 24
  Difference in the percentage of participants with SALT score less than or equal to 20 between ritlecitinib 100 mg once-daily (QD) versus placebo

SECONDARY OUTCOMES:
Percentage of participants with absolute SALT score less than or equal to 20 | Week 24
  Difference in the percentage of participants with SALT score less than or equal to 20 between ritlecitinib 50 mg QD versus placebo
Change from baseline in SALT score | Week 24
  Difference in the mean absolute change from baseline in SALT score between ritlecitinib 100 mg QD versus ritlecitinib 50 mg QD
EU Only: Percentage of participants with Patient Global Impression of Change (PGI-C) response, defined as a score of "moderately improved" or "greatly improved" | Week 24
  Difference in percentage of participants with PGI-C response between ritlecitinib 100 mg QD versus placebo and ritlecitinib 50 mg QD versus placebo
US Only: Percentage of participants with absolute SALT score less than or equal to 20 | Week 36
  Difference in the percentage of participants with SALT score less than or equal to 20 between ritlecitinib 100 mg QD versus placebo
Percentage of participants with absolute SALT score less than or equal to 20 | Baseline through Week 24
  Difference in the percentage of participants with SALT score less than or equal to 20 between ritlecitinib 100 mg QD versus ritlecitinib 50 mg QD
Percentage of participants with absolute SALT score less than or equal to 10 | Baseline through Week 24
  Difference in the percentage of participants with SALT score less than or equal to 10 between ritlecitinib 100 mg QD versus ritlecitinib 50 mg QD
Percentage of participants with absolute SALT score equal to 0 | Baseline through Week 24
  Difference in the percentage of participants with SALT score equal to 0 between ritlecitinib 100 mg QD versus ritlecitinib 50 mg QD
Change from baseline in SALT score | Baseline through Week 24
  Difference in the mean absolute change from baseline in SALT score between ritlecitinib 100 mg QD versus ritlecitinib 50 mg QD
Percentage of participants with EBA (Eyebrow Assessment) response, defined as at least a 2-grade improvement from baseline or a score of 3 (among participants without a normal EBA score at baseline) | Baseline through Week 24
  Difference in the percentage of participants with EBA response (among participants without a normal EBA score at baseline) between ritlecitinib 100 mg QD versus ritlecitinib 50 mg QD
Percentage of participants with ELA (Eyelash Assessment) response, defined as at least a 2-grade improvement from baseline or a score of 3 (among participants without a normal ELA score at baseline) | Baseline through Week 24
  Difference in the percentage of participants with ELA response (among participants without a normal ELA score at baseline) between ritlecitinib 100 mg QD versus ritlecitinib 50 mg QD
Percentage of participants with PGI-C response, defined as a score of "moderately improved" or "greatly improved" | Baseline through Week 24
  Difference in the percentage of participants with PGI-C response between ritlecitinib 100 mg QD versus ritlecitinib 50 mg QD
Percentage of participants with absolute SALT score less than or equal to 10 | Week 24
  Difference in the percentage of participants with SALT score less than or equal to 10 between ritlecitinib 100 mg QD versus placebo and ritlecitinib 50 mg QD versus placebo
Percentage of participants with EBA response, defined as at least a 2-grade improvement from baseline or a score of 3 (among participants without a normal EBA score at baseline) | Week 24
  Difference in the percentage of participants with EBA response (among participants without a normal EBA score at baseline) between ritlecitinib 100 mg QD versus placebo and ritlecitinib 50 mg QD versus placebo
Percentage of participants with ELA response, defined as at least a 2-grade improvement from baseline or a score of 3 (among participants without a normal ELA score at baseline) | Week 24
  Difference in the percentage of participants with ELA response (among participants without a normal ELA score at baseline) between ritlecitinib 100 mg QD versus placebo and ritlecitinib 50 mg QD versus placebo
Percentage of participants with absolute SALT score less than or equal to 20 | Week 48
  Difference in the percentage of participants with SALT score less than or equal to 20 between ritlecitinib 50 mg non-responder (NR)-->ritlecitinib 100 mg QD versus ritlecitinib 50 mg NR-->ritlecitinib 50 mg QD
Percentage of participants with absolute SALT score less than or equal to 10 | Week 48
  Difference in the percentage of participants with SALT score less than or equal to 10 between ritlecitinib 50 mg NR-->ritlecitinib 100 mg QD versus ritlecitinib 50 mg NR-->ritlecitinib 50 mg QD
Change from Week 24 in SALT score | Week 48
  Difference in the mean absolute change from Week 24 in SALT score between ritlecitinib 50 mg NR-->ritlecitinib 100 mg QD versus ritlecitinib 50 mg NR-->ritlecitinib 50 mg QD
Percentage of participants with PGI-C response, defined as a score of "moderately improved" or "greatly improved" | Week 48
  Percentage of participants with PGI-C response between ritlecitinib 50 mg NR-->ritlecitinib 100 mg QD versus ritlecitinib 50 mg NR-->ritlecitinib 50 mg QD
Percentage of participants with absolute SALT score less than or equal to 20 | Week 24 through Week 48
  Percentage of participants with SALT score less than or equal to 20 for ritlecitinib 100 mg QD, ritlecitinib 50 mg responder (R)-->50 mg QD, ritlecitinib 50 mg NR-->50 mg QD, and ritlecitinib 50 mg NR-->100 mg QD
Percentage of participants with absolute SALT score less than or equal to 10 | Week 24 through Week 48
  Percentage of participants with SALT score less than or equal to 10 for ritlecitinib 100 mg QD, ritlecitinib 50 mg R-->50 mg QD, ritlecitinib 50 mg NR-->50 mg QD, and ritlecitinib 50 mg NR-->100 mg QD
Percentage of participants with SALT score equal to 0 | Week 24 through Week 48
  Percentage of participants with SALT score equal to 0 for ritlecitinib 100 mg QD, ritlecitinib 50 mg R-->50 mg QD, ritlecitinib 50 mg NR-->50 mg QD, and ritlecitinib 50 mg NR-->100 mg QD
Change from Week 24 in SALT score | Week 24 through Week 48
  Mean absolute change from Week 24 in SALT score for ritlecitinib 100 mg QD, ritlecitinib 50 mg R-->50 mg QD, ritlecitinib 50 mg NR-->50 mg QD, and ritlecitinib 50 mg NR-->100 mg QD
Percentage of participants with EBA response, defined as at least a 2-grade improvement from baseline or a score of 3 (among participants without a normal EBA score at baseline) | Week 24 through Week 48
  Percentage of participants with EBA response for ritlecitinib 100 mg QD, ritlecitinib 50 mg R-->50 mg QD, ritlecitinib 50 mg NR-->50 mg QD, and ritlecitinib 50 mg NR-->100 mg QD
Percentage of participants with ELA response, defined as at least a 2-grade improvement from baseline or a score of 3 (among participants without a normal ELA score at baseline) | Week 24 through Week 48
  Percentage of participants with ELA response for ritlecitinib 100 mg QD, ritlecitinib 50 mg R-->50 mg QD, ritlecitinib 50 mg NR-->50 mg QD, and ritlecitinib 50 mg NR-->100 mg QD
Percentage of participants with PGI-C response, defined as a score of "moderately improved" or "greatly improved" | Week 24 through Week 48
  Percentage of participants with PGI-C response for ritlecitinib 100 mg QD, ritlecitinib 50 mg R-->50 mg QD, ritlecitinib 50 mg NR-->50 mg QD, and ritlecitinib 50 mg NR-->100 mg QD

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (113):
- United States (45):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Doc1 Healthcare Systems, Brea, California
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Marvel Clinical Research, Huntington Beach, California
  - Southern California Clinical Research, Santa Ana, California
  - Brett King MD, LLC, Fairfield, Connecticut
  - Alliance for Multispecialty Research, LLC, Fort Myers, Florida
  - Robert B. Pritt, DO, PA, Fort Myers, Florida
  - Solutions Through Advanced Research, Jacksonville, Florida
  - Pediatric Skin Research, Miami, Florida
  - Skin Research of South Florida, Miami, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Olympian Clinical Research - Tampa - Memorial Highway, Tampa, Florida
  - Endeavor Health, Skokie, Illinois
  - Indiana University Health University Hospital Adult Outpatient Center, Indianapolis, Indiana
  - Indiana University School of Medicine - Indiana CTSI Clinical Research Center, Indianapolis, Indiana
  - Sidney & Lois Eskenazi Health Center, Indianapolis, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Callender Center for Clinical Research, Glenn Dale, Maryland
  - Dermatology and Skin Cancer Specialists, LLC, Rockville, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Revival Research Institute, LLC, Troy, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Clinical & Translational Research Center (CTRC), Chapel Hill, North Carolina
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - Bexley Dermatology Research, Bexley, Ohio
  - Apex Clinical Research Center - Canton, Canton, Ohio
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Oregon Medical Research Center, Portland, Oregon
  - Northwest Dermatology Institute, Portland, Oregon
  - NW Dermatology Institute, Portland, Oregon
  - Dermatology Associates of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - Alliance for Multispecialty Research, LLC, Myrtle Beach, South Carolina
  - Arlington Research Center, Arlington, Texas
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Center for Clinical Studies - Clear Lake, Webster, Texas
  - AMR Clinical, Layton, Utah
  - University of Utah, Murray, Utah
  - Dermatology Specialists of Spokane, Spokane, Washington
  - Principle Research Solutions, Spokane, Washington
- Canada (16):
  - CaRe Clinic, Red Deer, Alberta
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Guelph Dermatology Research, Guelph, Ontario
  - DermEffects, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - Ryan Clinical Research Inc., Newmarket, Ontario
  - The Centre for Clinical Trials, Oakville, Ontario
  - JRB Research Inc., Ottawa, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - Research Toronto, Toronto, Ontario
  - Centre de Recherche Saint-Louis, Montreal, Quebec
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Saint-Louis, Sherbrooke, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain, Québec
  - Centre de Recherche Saint-Louis inc., Québec
- China (16):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Children's hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - 2nd Affiliated Hospital Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangxi Provincial Children's Hospital, Nanchang, Other
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Chengdu Second Municipal People's Hospital, Chengdu, Sichuan
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou Third Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Friendship hospital, Capital Medical University, Beijing
  - Nanjing Medical University (NMU) - Jiangsu Province Hospital, Nanjing
  - Shanghai Children's Hospital, Shanghai
- Kozni ambulance Fialova s.r.o, Prague, Praha 6, Czechia
- Japan (8):
  - Kurume University Hospital, Kurume, Fukuoka
  - Tohoku University Hospital, Sendai, Miyagi
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Juntendo Tokyo Koto Geriatric Medical Center, Koto-ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Niigata University Medical & Dental Hospital, Niigata
  - Osaka Metropolitan University Hospital, Osaka
- Poland (10):
  - Twoja Przychodnia PCM, Poznan, Greater Poland Voivodeship
  - Specjalistyczny Gabinet Dermatologiczny Aplikacyjno-Badawczy, Marek Brzewski, Paweł Brzewski spółka, Krakow, Lesser Poland Voivodeship
  - Cityclinic Przychodnia Lekarsko-Psychologiczna Matusiak Spółka Partnerska, Wroclaw, Lower Silesian Voivodeship
  - DERMEDIC Iwona Zdybska, Lublin, Lublin Voivodeship
  - Twoja Przychodnia NCM, Nowa Sól, Lubusz Voivodeship
  - Klinika Osipowicz & Turkowski, Warsaw, Masovian Voivodeship
  - Royalderm Agnieszka Nawrocka, Warsaw, Masovian Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne Angelius Provita, Katowice, Silesian Voivodeship
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin, West Pomeranian Voivodeship
- South Korea (10):
  - Dankook University Hospital, Cheonan-si, Chungcheongnam-do [chungnam]
  - Jeonbuk National University Hospital, Jeonju, Jeonrabugdo
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Pusan National University Hospital, Busan, Pusan-kwangyǒkshi
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Konkuk University Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Kyung Hee University Hospital at Gangdong, Seoul, Seoul-teukbyeolsi [seoul]
  - Boramae Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Kyungpook National University Hospital, Junggu, Taegu-kwangyǒkshi
- Spain (2):
  - AUDIKA, Córdoba, Andalusia
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
- Taiwan (5):
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist, Kaohsiung
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] King B, McMichael A, Sinclair R, Vano-Galvan S, Wolk R, Woodworth D, Soma K, Robbana F, Lejeune A, Napatalung L, Law E, Wajsbrot D, Wang C, Roychoudhury S. Rationale and Design of a Novel, Phase 3, External and Synthetic Placebo-Controlled Clinical Trial of Ritlecitinib 50 mg and 100 mg for Alopecia Areata. Dermatol Ther (Heidelb). 2025 Dec;15(12):3793-3803. doi: 10.1007/s13555-025-01543-7. Epub 2025 Oct 14. PMID 41083802
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981094
- See also: See if you/your child may be eligible for this clinical trial — https://www.allegro100clinicaltrial.com